CLINICAL TRIAL: NCT02751658
Title: Pathobiomes Training in the Care of Water Sources and Dynamics of Water-borne Pathogens Involved in Healthcare Associated Infections
Brief Title: Tap to "Tap", Pathobiome Associates Health Care
Acronym: TapPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9648
Record Dates: First submitted 2016-03-04; First posted 2016-04-26 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Otorhinolaryngologic Diseases
MeSH Terms: conditions — Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients in the Otorhinolaryngology (Other): patients in the Otorhinolaryngology department realization of a levy into the mouth swab on the day of admission to hospital and the day of release
  Interventions: Other: mouth swab

INTERVENTIONS:
Other: mouth swab — Levy to make inside of the mouth with a swab on the day of admission to hospital and the day of release at the patients in the Otorhinolaryngology

SUMMARY:
The bacteria live in community and in some cases it is the combination of several microorganisms that facilitates transmission and pathogenicity. The concept of pathobiome follows from this finding. Investigators hypothesize that the microbial community water point is a pathobiome influencing installation and transmission of pathogens associated with care

DETAILED DESCRIPTION:
Goals :

Key: To study the impact of bacterial communities on the risk of transmission of waterborne pathogenic bacterium Pseudomonas aeruginosa in patients hospitalized from a contaminated water source by this bacterium.

secondary:

1. Assess the role of communities on installing the water points in P. aeruginosa by comparing contaminated and uncontaminated water sources.
2. To evaluate the effect of the quality of water and the conditions of use of water points network on the composition of bacterial communities associated or not with P. aeruginosa.

Experimental Study conducted from 6 points of water, contaminated deliberately experimental backs onto the project to assess conventional and alternative measures decontamination network and water points

ELIGIBILITY:
Inclusion Criteria:

* Patients in the Otorhinolaryngology department

Exclusion Criteria:

* Immunocompromised patients
* Patient Opposition to enter the research protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Presence of Pseudomonas aeruginosa | Entrance hospitalization (Day 1)
  The presence of Pseudomonas aeruginosa will be made from a buccal swab in all patients admitted to the hospital entrance.
  Mark of Pseudomonas aeruginosa will be done with and without trypticase soy broth enrichment and isolation on selective agar cetrimide Pseudomonas aeruginosa . The enrichment will detect a port at very low inoculum knowing that the purpose of the analysis is to detect passing of Pseudomonas aeruginosa from the environment to the patient regardless of the associated infectivity. The identification of certainty will be carried out by MALDI-TOF. If several morphotypes are visualized on agar Cetrimide they will all be identified and kept under custody broth at -20 ° C.

SECONDARY OUTCOMES:
Presence of infection with Pseudomonas aeruginosa | Exit hospitalization (Day 10)
  The presence of Pseudomonas aeruginosa will be made from a buccal swab in all patients exit hospitalization.
  Mark of Pseudomonas aeruginosa will be done with and without trypticase soy broth enrichment and isolation on selective agar cetrimide Pseudomonas aeruginosa . The enrichment will detect a port at very low inoculum knowing that the purpose of the analysis is to detect passing of Pseudomonas aeruginosa from the environment to the patient regardless of the associated infectivity. The identification of certainty will be carried out by MALDI-TOF. If several morphotypes are visualized on agar Cetrimide they will all be identified and kept under custody broth at -20 ° C.

CONTACTS AND LOCATIONS:
Overall Officials: Sara ROMANO-BERTRAND, MCU-PH, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Benigno V, Carraro N, Sarton-Loheac G, Romano-Bertrand S, Blanc DS, van der Meer JR. Diversity and evolution of an abundant ICEclc family of integrative and conjugative elements in Pseudomonas aeruginosa. mSphere. 2023 Dec 20;8(6):e0051723. doi: 10.1128/msphere.00517-23. Epub 2023 Oct 30. PMID 37902330
- [Derived] Virieux-Petit M, Hammer-Dedet F, Aujoulat F, Jumas-Bilak E, Romano-Bertrand S. From Copper Tolerance to Resistance in Pseudomonas aeruginosa towards Patho-Adaptation and Hospital Success. Genes (Basel). 2022 Feb 4;13(2):301. doi: 10.3390/genes13020301. PMID 35205346